CLINICAL TRIAL: NCT03395743
Title: Expanded Access Program for AB-PA01, an Investigational Anti-Pseudomonas Aeruginosa Bacteriophage Therapeutic, for the Treatment of Individual Patients With Serious or Immediately Life-threatening Infections Caused by Pseudomonas Aeruginosa
Brief Title: Individual Patient Expanded Access for AB-PA01, an Investigational Anti-Pseudomonas Aeruginosa Bacteriophage Therapeutic
Status: No longer available | Type: Expanded Access
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-PA01-EAP01
Record Dates: First submitted 2017-12-19; First posted 2018-01-10 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: AB-PA01 — AB-PA01 is an investigational bacteriophage therapeutic for treatment of Pseudomonas aeruginosa infections

SUMMARY:
The purpose of the expanded access program is to allow physicians to provide treatment with investigational drug, AB-PA01, for patients with serious or immediately life-threatening Pseudomonas aeruginosa infections, for which no alternative treatment(s) are currently available, and who meet the criteria for treatment under FDA's Expanded Access regulations and criteria set forth by AmpliPhi Biosciences Corporation.

To be considered for expanded access, the request should be submitted to AmpliPhi by a qualified and licensed physician with expertise and facilities appropriate for the administration of the investigational medicine. Treating physicians should contact AmpliPhi by emailing expandedaccess@ampliphibio.com with "Expanded Access Request" in the subject line, and include in the email the treating physicians name, organization/hospital/institution, physical address, email address, telephone number, and a brief description of the indication/condition.

Any approval of expanded access to investigational medicine must always comply with the applicable laws and regulations.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult